CLINICAL TRIAL: NCT04913948
Title: Assessing the Mother-to-infant Transmission Capabilities of COVID-19 Infection Among Pregnant Women in Ontario, Canada
Acronym: COPE
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: CTO 2168
Record Dates: First submitted 2021-03-03; First posted 2021-06-04 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: SARS-CoV-2; Covid19; Corona Virus Infection; Infectious Disease Transmission, Vertical; Pregnancy
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Should residual samples (i.e. maternal serum, umbilical cord serum, amniotic fluid, breast milk, placental tissue [frozen and fixed]) remain after the purposes of the primary outcomes, samples will be retained for 10 years for future, related REB approved studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant: Pregnant women with confirmed COVID-19 at any point during pregnancy or suspected (as identified at local hospital) of COVID-19 at time of delivery, who will be delivering at a participating hospital
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
In order to assess the mother-to-infant and potential vertical transmission of SARS-CoV-2 infection in pregnant women, maternal and neonatal biological samples were prospectively collected from women with confirmed or suspected COVID-19 at participating hospitals. Samples were be tested for the SARS-CoV-2 serology and presence of SARS-CoV-2 RNA.

Outcomes for the study objective will be ascertained through the collection and testing of biological samples from the mother and/or infant. Specifically the investigators will:

1. Assess maternal nasopharyngeal or oropharyngeal swab, vaginal mucosa, ano-rectal swab, amniotic fluid, placenta (including subamniotic swab), breastmilk, cord blood and neonatal nasopharyngeal swab for RNA particles of coronavirus, by ddPCR.
2. Assess maternal serum for anti-coronavirus antibodies, by immunoassay.
3. Examine the impact of coronavirus on the neonate with respect to serology and viral load, in addition to placenta pathology findings and ddPCR.
4. Assess vertical transmission and the effect of coronavirus through placental pathology examination using placental pathology synoptic report.

DETAILED DESCRIPTION:
Pregnant individuals with severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infection were more likely to experience greater disease severity and higher rates of hospitalization, intensive care unit (ICU) admission and death compared to their non-pregnant counterparts. Early pandemic data were limited to a few small case series and reports that failed to provide a clear understanding of the timing and likelihood of fetal/neonatal infection. Data now suggest that in utero, intrapartum and early postnatal transmission of SARS-CoV-2 to the fetus/neonate is rare (<5%) and predominantly associated with third trimester infections and severe disease presentation. A living systematic review and meta-analysis of 144 cohort studies found that the rate neonates/fetuses testing positive for SARS-CoV-2 by RT-PCR, having anti-SARS-CoV-2 IgM antibodies or both was 1.94% (95%CI 1.31%, 2.66%). However, tests for SARS-CoV-2 and anti-SARS-CoV-2 antibodies were limited during the earliest stages of the pandemic and relatively few of the included studies provided sufficient data on the timing of fetal/neonatal exposure, and the type and timing of tests performed.

Derivation of reliable risk estimates for perinatal transmission remains challenging due to significant heterogeneity across published studies regarding the types of tissues profiled, diagnostic methods used and availability of essential COVID-19 disease characteristics such as timing and severity of maternal infection. As variants of concern continue to emerge, more data are required to elucidate the circumstances in which SARS-CoV-2 infection is likely to be transmitted to the developing fetus/neonate. We sought to evaluate the rate of SARS-CoV-2 transmission from mother-to-neonate in a large multicenter cohort from Ontario and Quebec, Canada.

To address early pandemic challenges in characterizing perinatal infections, a prospective cohort study was conducted across 14 sites in Ontario and Quebec, Canada. Pregnant individuals who had received a diagnosis of SARS-CoV-2 infection in pregnancy were eligible. Sample collection at delivery included maternal samples (nasopharyngeal/oropharyngeal, vaginal and anorectal swabs; blood; breastmilk), newborn samples (nasopharyngeal swabs, cord blood, amniotic fluid), and placental samples (sub-amniotic swab, placental biopsies). Swab, amniotic fluid, placenta and breastmilk samples were analyzed for SARS-CoV-2 RNA by RT-qPCR. Blood, breastmilk and amniotic fluid were assessed for anti-SARS-CoV-2 spike (S), receptor binding domain (RBD) and nucleocapsid (N) IgG, IgM and IgA.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with confirmed COVID-19 at any point during pregnancy or suspected COVID-19 at time of delivery (as identified at local hospital) , who will be delivering at a participating hospital in Ontario or Quebec

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women meeting the study eligibility criteria and delivering at a participating hospital within Ontario or Quebec will be recruited. Hospitals within the COPE Network include both Level II and III hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darine El-Chaar, MD, MSc, Principal Investigator — The Ottawa Hospital
Locations (12):
- Canada (12):
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - London Health Sciences, London, Ontario
  - North York General Hospital, North York, Ontario
  - Humber River Hospital, North York, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Hôpital Montfort, Ottawa, Ontario
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
IPD that underlie the results reported in this article, after deidentification, will be made available to other researchers upon request.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pregnant
Started | 246
Completed | 242
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Sample processing issues | 1
Not completed — Suspected to have COVID-19 at the time of delivery but was found to be negative upon RT-PCR testing | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pregnant
Number analyzed (Participants) | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 242
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 69
  Asian | 35
  Black | 43
  Other/Unknown/Mixed ethnicity | 20
  Missing | 75
Neighbourhood family income quintile [Count of Participants; unit: Participants]
  Quintile 1 (lowest) | 60
  Quintile 2 | 48
  Quintile 3 | 40
  Quintile 4 | 34
  Quintile 5 | 28
  Missing | 32
Pre-pregnancy BMI [Count of Participants; unit: Participants] — Body mass index before pregnancy.
  Participants
    <18.5 | 6
    18.5 to <25 | 93
    25 to >30 | 68
    >=30 | 67
    Missing | 8
Gestational weight gain [Count of Participants; unit: Participants] — Based on 2009 Institute of Medicine recommendations, whereby recommended gestational weight gain (lb) is based on pre-pregnancy BMI (kg/m2) as follows:
  28lb-40lb for pre-pregnancy BMI <18.5 kg/m2 25-35lb for pre-pregnancy BMI 18.5-24.9 kg/m2 15-25lb for pre-pregnancy BMI 25.0-29.9 kg/m2 11-20lb for pre-pregnancy BMI ≥30 kg/m2 Weight gain within recommended ranges are considered optimal.
  Participants
    Less than recommended | 50
    Within recommended range | 43
    More than recommended | 112
    Missing | 37
Parity [Count of Participants; unit: Participants] — Where nulliparous refers to an individual who has never given birth; primiparous refers to an individual who has given birth once; multiparous refers to an individual who has given birth more than once.
  Participants
    Nulliparous | 50
    Primiparous | 43
    Multiparous | 112
    Missing | 37

OUTCOME MEASURES:

1. Primary Outcome: Rate of Perinatal Transmission of SARS-CoV-2
Description: Evidence of SARS-CoV-2 RNA or antibodies against SARS-CoV-2 from a sterile (amniotic fluid) or non-sterile sample (nasopharyngeal swab sample, placental tissue, subamniotic swab or by cord blood serology [for IgM or IgA]) collected during the maternal hospital admission for delivery (specific time frame varied per participant).
Time Frame: During the delivery admission
Population: The rate of perinatal transmission of SARS-CoV-2 was estimated based on one or more positive test results by RT-PCR for SARS-CoV-2 from a sterile (amniotic fluid) or non-sterile sample (nasopharyngeal swab sample, placental tissue, subamniotic swab) or by cord blood serology (for IgM or IgA). A total of 227 participant provided the appropriate samples for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Pregnant
Number analyzed (Participants) | 227
percentage of participants | 12.3

2. Primary Outcome: Rate of Intrauterine Transmission of SARS-CoV-2
Description: Evidence of SARS-CoV-2 RNA or antibodies against SARS-CoV-2 in fetal tissues (i.e., amniotic fluid, placental tissue, sub-amniotic swab, cord blood) collected during maternal hospital admission for delivery (specific time frame varied per participant). Evidence of intrauterine transmission was determined using RT-PCR and serological analysis.
Time Frame: During the delivery admission
Measure: Number; unit: percentage of participants
Arm/Group | Pregnant
Number analyzed (Participants) | 227
percentage of participants | 4.4

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 6 weeks postpartum
Arm/Group | Pregnant
All-Cause Mortality (participants affected / at risk) | 0/242
Serious Adverse Events (participants affected / at risk) | 0/242
Other Adverse Events (participants affected / at risk) | 0/242

LIMITATIONS AND CAVEATS:
First, this was a convenience sample of individuals from Ontario and Quebec. Second, our ability to collect all samples from all participants was affected by local resources for safe sample collection, processing, storage, and patient preferences. Finally, our findings may not be generalizable to settings where SARS-CoV-2 community transmission rates and related outcomes varied significantly over the course of the pandemic, by variant and by local public health policies and practices.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT04913948/Prot_SAP_000.pdf